CLINICAL TRIAL: NCT02372266
Title: A Randomized Controlled Trial to Assess the Safety and Cost-Effectiveness of Early Maternal Newborn Infant Discharge
Brief Title: Safety and Cost-Effectiveness of Early Maternal Newborn Infant Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Responsible Party: Principal Investigator, William H. Barth, Jr., M.D., Col(ret), USAF, MC, Chairman, Department of Obstetrics and Gynecology, 59th Medical Wing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGO 96-042; DI950076 (Other Grant/Funding Number: Department of Defense Women's Health Intramural Research); FWH19960042H (Other: Wilford Hall Medical Center)
Record Dates: First submitted 2015-02-03; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Pregnancy
Keywords: Infant, Newborn; hospital discharge; Early newborn discharge; Newborn length of stay; Maternity length of stay

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Discharge Group (Experimental): If safety criteria were met, women and infants were discharged home from the hospital at 12 to 24 hours after delivery with a planned home health visit within 48 hours of the discharge.
  Interventions: Other: Early Maternal-Newborn Infant Discharge
- Routine Stay Group (Active Comparator): Women and newborns were discharged no sooner than 48 hours after delivery and could stay voluntarily up to 72 hours.
  Interventions: Other: Routine discharge

INTERVENTIONS:
Other: Early Maternal-Newborn Infant Discharge — Discharge from the hospital between 12-24 hours of life
  Arms: Early Discharge Group
Other: Routine discharge — Discharge of the mother and newborn 2 to 3 days after delivery
  Arms: Routine Stay Group

SUMMARY:
To determine the effect of a policy of early maternal-newborn infant discharge (12-24 hours) with a home visit on admission to the Level II/III nursery and hospital admissions and readmissions.

DETAILED DESCRIPTION:
This is a randomized controlled trial designed to assess the safety of a policy of early maternal newborn infant discharge compared to a policy of routine discharge 2 to 3 days after delivery. The primary outcome is newborn admissions to the Level II or Level III neonatal care unit or hospital within three days of delivery. Secondary outcomes included admissions and readmissions at 2 weeks, 6 weeks and 6 months following delivery, maternal satisfaction with length of stay and overall birthing experience, lactation continuation rates, maternal anxiety, depression, confidence and family functioning. We applied the American Academy of Pediatrics criteria for early newborn discharge, but planned the analysis by intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women enrolling for obstetric care at a large military academic health center

Exclusion Criteria:

* Planning a move from the area before delivery
* Multiple gestations
* Pre-existing maternal diabetes
* Maternal chronic hypertension
* Maternal age < 18

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2223 (Actual)
Dates: Start 1997-04; Primary Completion 2001-01 (Actual); Study Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
Admission to the Level II/III neonatal care unit or hospital | 72 hours
  All admissions to the Level II/III neonatal care unit following delivery

SECONDARY OUTCOMES:
Emergency department visits, clinic visits, or hospital admissions | 72 hours
  Any unplanned pediatric visit to an emergency room, clinic or a hospital admission
Emergency department visits, clinic visits, or hospital admissions | 14 days
  Any unplanned pediatric visit to an emergency room, clinic or a hospital admission
Emergency department visits, clinic visits, or hospital admissions | 8 weeks
  Any unplanned pediatric visit to an emergency room, clinic or a hospital admission
Emergency department visits, clinic visits, or hospital admissions | 6 months
  Any unplanned pediatric visit to an emergency room, clinic or a hospital admission
Breastfeeding score (5 point Likert scale) | At discharge (12 to 72 hours after delivery)
  5 point Likert scale: Only breast, mostly breast, 50/50, mostly bottle, only bottle
Breastfeeding score (5 point Likert scale) | 14 days
  5 point Likert scale: Only breast, mostly breast, 50/50, mostly bottle, only bottle
Breastfeeding score (5 point Likert scale) | 8 weeks
  5 point Likert scale: Only breast, mostly breast, 50/50, mostly bottle, only bottle
Breastfeeding score (5 point Likert scale) | 6 months
  5 point Likert scale: Only breast, mostly breast, 50/50, mostly bottle, only bottle
Maternal anxiety (State/Trait Anxiety Inventory) | At discharge (12 to 72 hours after delivery)
Maternal anxiety (State/Trait Anxiety Inventory) | 14 days
  State/Trait Anxiety Inventory
Maternal depression (Generalized Contentment Scale) | At discharge (12 to 72 hours after delivery)
  Generalized Contentment Scale
Maternal depression (Generalized Contentment Scale) | 14 days
  Generalized Contentment Scale
Maternal confidence (Confidence on a Likert scale) | At discharge (12 to 72 hours after delivery)
  Confidence on a Likert scale
Maternal confidence (Confidence on a Likert scale) | 14 days
  Confidence on a Likert scale
Maternal satisfaction with length of stay (Likert scale) | At discharge (12 to 72 hours after delivery)
  Satisfaction with length of stay on a Likert scale
Maternal satisfaction with length of stay (Likert scale) | 14 days
  Satisfaction with length of stay on a Likert scale
Maternal satisfaction with overall experience (Likert scale) | At discharge (12 to 72 hours after delivery)
  Satisfaction with overall childbirth experience on a Likert scale
Maternal satisfaction with overall experience (Likert scale) | 14 days
  Satisfaction with overall childbirth experience on a Likert scale
Admission to the Level II/III neonatal care unit or hospital | 14 days
  All admissions to the Level II/III neonatal care unit following delivery
Admission to the Level II/III neonatal care unit or hospital | 8 weeks
  All admissions to the Level II/III neonatal care unit following delivery
Admission to the Level II/III neonatal care unit or hospital | 6 months
  All admissions to the Level II/III neonatal care unit following delivery

CONTACTS AND LOCATIONS:
Overall Officials: William H Barth, MD, Principal Investigator — Massachusetts General Hospital